CLINICAL TRIAL: NCT04831905
Title: Etude de faisabilité de de tolérance d'un Traitement Focal Transrectal Par Micro-ondes de la Tumeur Index Des Patients Ayant un Cancer de la Prostate - FOSTINE 1b
Brief Title: Micro-wave Ablation Under Organ-based Tracking in Patients With Prostate Cancer - FOSTINE
Acronym: FOSTINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Collaborators: Koelis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOSTINE
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Focal Treatment for Prostate Cancer
Keywords: prostate cancer; Focal treatment for prostate cancer; Focal treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Ablate and resect study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilote study (Experimental): Micro-wave ablation of index lesion identified on MRi on prostate cancer
  Interventions: Device: Micro-wave ablation

INTERVENTIONS:
Device: Micro-wave ablation — Micro-wave ablation

SUMMARY:
With the advent of multiparametric MRI (mpMRI), the concept of focal therapy continues to develop as a compromise between active surveillance and radical tratment. However, it must be combined with the most stringent quality control measures, such as exceptional Imaging, to allow close management of the index tumor. the choice of the energy is also crucial. Several have been tested such as HIFU, electroporation or cryotherapy. A new therapeutic alternative currently Under investigation resides in the use of microwaves delivered through a thin needle inserted precisely into the index lesion according to the same procedure as targeted biopsy under image fusion to induce coagulation necrosis and lead to the tumor destruction. Through an ablate, performed transrectally under real-time MRI/TRUS image registration and 3D mapping, in patients with localized prostate cancer (PCa).

DETAILED DESCRIPTION:
Patients with a detectable index lesion on mpMRI, PSA level <20 ng/mL and wishing to undergo a prostatectomy due to significant PCa on biopsy are elibible for this study approved by the Ethics Committee. Targeted biopsies of the index lesion are performed by using an ultrasound-MRI image fusion system with Organ based Tracking (OBT)-registration (Trinity*, KOELIS, France) to provide quality control. Targeted cores are analyzed intraoperatively with an extemporaneoux analyses. If positive, a targeted focal microwave ablation is achieved during the same session by a single 18G needle inserted transrectally Under sedation. Predictive ablation charts obtained with the 2.45 GHZ frequency microwave generator (TATO, Biomedical Srl, Italy) through ex vivo experiments were used to choose the duration and power of the treatment.

Treated patients are followed-up for 4 to 6 weeks and the planned radical prostatectomy is performed. All treated patients complete uroflowmetry test and questionnaires (IPSS, IPSS-QQL, IIEF-5, and MSHW-EJD-SF) befor, at 7 days and 1 month after the procedure. A mpMRI of the treated prostate is performed at 7 days after the ablation to identify the devascularized area, but also to verify that no organ at risk is affected by the microweve treatment. After radical prostatectomy, whole-mount histology serves to define the ablation boundaries and dimension in the prostate. It also allows to determine the impact of the use of microwaves on cancerous tissue. A total of 10 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with detectable index lesion on mpMRI, PSA level <20 ng/mL and wishing to undergo a prostatectomy due to significant PCA on biopsy.
* Life expectancy up to 10 years or plus.

Exclusion Criteria:

* Past history of prostate surgery or pelvic radiotherapy, prostatitis, extra-capsular extension on MRI or index lesion above 25 mm, distance between rectum and index lesion less than 5 mm.

Ages: 45 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Micro-wave ablation area | 6 weeks
  Tolerance and faisability of transerectal micro wave ablation of index lesion in prostate cancer.

SECONDARY OUTCOMES:
Micro-wave ablation area | 6 weeks
  MRI to identify the devascularized area at one week and ablation boundaries and dimensions in the prostate specimen after prostatectomy at one month.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
anonymising patients personal data for publications

REFERENCES:
- See also: Fusion device — https://koelis.com/en/